CLINICAL TRIAL: NCT05553587
Title: Perceived Changes in Symptom Burden and Physiological Effects of a Proprietary Phyto-therapeutic Preparation (Amara) in Patients With Functional Dyspepsia: Prospective Study as Investigator Initiated Trial (IIT)
Brief Title: Symptoms and Physiological Effects of Amara in Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mark Fox (Other)
Responsible Party: Sponsor-Investigator, Mark Fox, Prof. Dr. med., Klinik Arlesheim
Organization: Klinik Arlesheim (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amara-KLA-01-22
Record Dates: First submitted 2022-06-14; First posted 2022-09-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Dyspepsia
Keywords: Phytotherapy; Gastric Emptying; Gastric Sensation; Clinical Outcomes Research
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: prospective, open label, non-randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amara Drops (Experimental): Phytopharmaceutical / therapeutic intervention
  Interventions: Drug: Amara drops

INTERVENTIONS:
Drug: Amara drops — The investigational drug is approved with a reduced dossier without indication according to Art. 25 para. 1 KPAV (SR 812.212.24). This study follows the indication text licensed by Swissmedic: "… Weleda Amara-Drops can be used for digestive complaints such as heartburn, flatulence and bloating after meals, to stimulate the bile flow and for loss of appetite and nausea. The effect of Weleda Amara drops is based on a balanced mixture of medicinal plants with tonic (invigorating) and aromatic bitter substances, which are suitable for stimulating digestion." Further, no side effects have been reported in past studies so far. All these reasons lead us to the conclusion that this study is only associated with minimal risks and should be classified in risk category A.

SUMMARY:
The primary aim of this investigator-initiated, prospective, open-label study is to assess perceived changes in symptom burden reported by in patients with functional dyspepsia treated with Amara. Additionally, the physiological effects of Amara on gastric motor and sensory function will be assessed using validated methods.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) with postprandial distress is a common functional gastrointestinal (GI) disorder characterized by the occurrence of epigastric symptoms such as early satiety (fullness), nausea and upper abdominal pain after meals at least twice a week over at least six months (Rome IV criteria). By definition, no structural disease is found on routine endoscopy or imaging studies. Instead, symptoms are thought to be related to abnormal gastrointestinal motility (e.g., impaired gastric relaxation, abnormal emptying) and increased sensitivity to gastric distension and the digestive process.

Epidemiological studies report a 10-30% prevalence of functional dyspepsia (FD) worldwide. When dyspeptic symptoms are short in duration and relatively mild, many patients wish to self-manage with dietary adaptation and /or over the counter (OTC) preparations. Others report high rates of intolerance to prescription medications. In these patients complementary and alternative medicines (CAM) based on natural products, such as plant-based "phytotherapy", are particularly appealing. Several herbal therapies for functional dyspepsia have been tested in randomized clinical studies. These include phytochemicals such as peppermint oil that inhibits smooth muscle contraction by direct blockade of calcium channels and other effects, deglycyrrhizinated licorice that increases gastric mucus secretion and may enhance mucosal protection and other preparations that combine multiple herbal products with the intention of inducing synergistic effects that promote normal digestive function. For example, a meta-analysis of 3 double blind RCTs provided evidence that STW-5 (Iberogast, Bayer) is more effective than placebo in the Treatment of dyspeptic symptoms.

Amara tincture (Weleda, Arlesheim, Switzerland) is a proprietary preparation used for many decades in complementary medicine that is marketed for the treatment of functional digestive disorders. Patients take 10-20 drops before meals to relieve loss of appetite, bloating, nausea, and other dyspeptic symptoms. These bitter substances are thought to promote digestion and relieve symptoms by stimulating the secretion of gastric and pancreatic enzymes, upper gastrointestinal motility and gastric emptying. These prokinetic effects may be therapeutic in patients with functional dyspepsia because there is an association between optimally measured delayed gastric emptying (GE) and upper gastrointestinal symptoms. To date, the effect of Amara has not been subjected to pre-clinical or clinical studies.

The primary aim of this investigator-initiated, prospective, open-label pilot therapeutic study is to assess perceived changes in symptom burden reported by in patients with functional dyspepsia treated with Amara. Additionally, the physiological effects of Amara on gastric motor and sensory function will be assessed using validated methods (Nutrient drink test followed by 13C gastric emptying study using the 400ml Nottingham Test Meal)

A prospective, open label, non-randomized study will assess (i) Perceived changes in symptom burden reported by patients during regular intake of 10-20 Amara Drops before main meals using the validated Leuven Dyspepsia Score.

(ii) Physiological effects of 20 drops Amara tincture on gastric emptying using the 400ml Nottingham Test Meal with non-radioactive 13C-acetate breath test and concurrent assessment of filling sensation and dyspeptic symptoms by Visual Analogue Scores (VAS).

Individuals that fulfill the diagnostic criteria for functional dyspepsia with postprandial distress syndrome according to the Rome IV criteria will be recruited. At the first study visit (Study Visit #1), Symptom questionnaires and other questionnaires to assess general gastroenterological health and psychiatric well-being will be completed at the time of recruitment. This data will be collected using an on-line application. Additionally, the Lüscher Color Test (LCT) will be performed. This non-verbal, non-written test has been developed to assess patient's personality and psychiatric state. This could be of interest in patients with disorders of brain-gut interaction that may not admit to the role of central factors in their illness.

Eligible patients will have no clinically relevant medical co-morbidity or previous gastrointestinal surgery and must have had a normal upper gastrointestinal pan-endoscopy in the previous 3 years. If not known, Helicobacter pylori status will be assessed by 13C-urea breath test (endoscopy not required). At this time, gastric function will be assessed by 13C-breath test measurements with concurrent assessment of visceral sensitivity after ingestion of a validated 400ml liquid "Nottingham Test Meal".

The LCT will be repeated at the second study visit (Study Visit #2), following a 2-4 week run-in period (no new treatments during this period). At this time, gastric function will be assessed again by 13C-breath test measurements with concurrent assessment of visceral sensitivity after ingestion of a validated 400ml liquid "Nottingham Test Meal (assess reproducibility)".

Amara Drops will be dispensed with 10-20 drops (0.25-0.50ml) taken three times a day prior to meals for 4 weeks. The patients are free to vary the dose between these limits as considered appropriate. The amount taken will be monitored by checking the volume remaining in the bottle at the end of the 4-week intervention. The presence and severity of dyspeptic symptoms and any side effects will be reported every day using an on-line application downloaded on the patient's smart phone (an electronic reminder will be sent at 21:00 every day).

At the end of the study period (Study Visit #3) the questionnaires including LCT and the 13C-breath test measurement with concurrent assessment of visceral sensitivity will be repeated on treatment. Additionally, the patients will be asked if their global satisfaction was better on Amara treatment, whether they wish to continue treatment and /or recommend the treatment to others with similar symptoms. Questionnaires and diary entries on side effects are also available as paper version.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred by their treating physician to the Center for integrative Gastroenterology at the Clinic Arlesheim
* Age over 18 years and ≦75 years of age
* Patients with Diagnosis of Functional Dyspepsia with Postprandial Distress (Rome IV criteria) with Leuven Dyspepsia Score "at least moderate" severity (>=10/20)
* Signed informed consent
* No change in medical treatment during the previous 1 month (e.g., proton pump inhibitor, antidepressants) during the last one month or for the duration of the period
* Good German knowledge (at least level B2 from Common European Framework of Reference for Languages)

Exclusion Criteria:

* Acute life-threatening conditions
* Withdrawal of informed consent
* Clinically relevant psychiatric comorbidity (HADS score >11)
* Advanced liver (Child score > 6) or kidney disease (GFR < 60)
* History of abdominal surgery except appendectomy
* Allergy to any component of Amara
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Dyspeptic Symptoms | 4 weeks (baseline and after intervention)
  The primary outcome will be the perceived change of dyspeptic symptoms assessed by the Leuven Dyspepsia Questionnaire (LDQ) between visit 2 (off treatment) and 3 (on treatment). It addresses 8 items distributed over five domains. The domains cover a range from 0 (none or absent) to 4(very severe) and assess symptom severity over the preceding 2 weeks. Higher total scores indicate more severe dyspeptic symptoms. The overall score ranges from 0-20 with standardized cut-offs: 0-5, normal to minimal dyspepsia; 6-10, mild dyspepsia; 10-15, moderate dyspepsia; 15-20, severe dyspepsia.

SECONDARY OUTCOMES:
Gastric Emptying | 4 weeks (baseline and after intervention)
  Change in gastric emptying as assessed by 13C Acetate Breath Test before and after 4 week Treatment with Amara (drug taken before test meal)
Visceral Sensitivity | 4 weeks (baseline and after intervention)
  Change in Gastric Filling Sensation and Dyspeptic Symptoms as assessed by Nutrient Drink Test (400ml Nottingham Test Meal) before and after 4 week Treatment with Amara (drug taken before test meal).
Reflux disease questionnaire (RDQ) | 4 weeks (baseline and after intervention)
  The RDQ ist a six item questionnaire to obtain information on the current frequency of reflux symptoms (heartburn, regurgitation and dyspepsia). Each item covers a range from 0-3 (never, 1 day, 2-3 days, 4-7 days) representing the frequency of the symptoms in the past seven days.
Irritable Bowel Syndrome - Severity Scoring System (IBS-SSS) | 4 weeks (baseline and after intervention)
  IBS-SSS is a five-item questionnaire measuring frequency and intensity of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and the interference of IBS with daily life, scoring from 0 to 100. Higher scores indicate more severe symptoms (mild 75-174, moderate 175-299, severe >300).

OTHER OUTCOMES:
The validity of the Lüscher Colour Test (LCT) | 4 weeks (baseline and after intervention)
  This will include face validity (debriefing session), construct validity (comparison with validated questionnaires assessing psychological patient related outcome measures), reproducibility (test re-test validity before and after run-in period), and internal consistency. Sensitivity of LCT to any change in dyspeptic symptoms, psychological or physiological state that occurs during the treatment study will also be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fox, MD MA, Principal Investigator — Lead Physician
Locations (1):
- Klinik Arlesheim, Arlesheim, Basel-Landschaft, Switzerland

DOCUMENTS (1):
  • Study Protocol (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT05553587/Prot_000.pdf